CLINICAL TRIAL: NCT05013086
Title: Therapeutic Efficiency and Response to 177Lu-AB-3PRGD2 in Patients With Integrin αVβ3 Positive Tumors
Brief Title: 177Lu-AB-3PRGD2 in Patients With Integrin αVβ3 Positive Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PekingUMCH AB-3PRGD2
Record Dates: First submitted 2021-08-13; First posted 2021-08-19 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Integrin αVβ3 Positive Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1.48 GBq of 177Lu-AB-3PRGD2 (Experimental): The patients were intravenously injected with the dose about 1.48GBq (40 mCi) of 177Lu-AB-3PRGD2 and underwent 68Ga-RGD PET/CT scans before and after the treatment.
  Interventions: Drug: 1.48 GBq of 177Lu-AB-3PRGD2

INTERVENTIONS:
Drug: 1.48 GBq of 177Lu-AB-3PRGD2 — accepted intravenous injection of 177Lu-AB-3PRGD2

SUMMARY:
This is an open-label, non-controlled, non-randomized study to assess the safety and measure image-based absorbed dose of 177Lu-AB-3PRGD2 in patients with Integrin αVβ3 positive tumors who will undergo radioliagnd therapy using 177Lu-AB-3PRGD2.

DETAILED DESCRIPTION:
Integrin αvβ3 is highly expressed in some tumor cells and neovascularization, which is an ideal target for diagnosis and treatment of Integrin αVβ3 positive tumors. 177Lu-AB-3PRGD2, is a kind of new drug based on independent research and development in China, provide an effective target for the treatment of Integrin αVβ3 positive tumors. All patients underwent whole-body 68Ga-RGD PET/CT for selection and accepted intravenous injection with single dose 1.48 GBq (40 mCi) of 177Lu-AB-3PRGD2 within one week. 1-2 ml venous blood was collected at 5min, 3h, 24h, 72h and 168h after administration to detect radioactivity count, respectively. Then monitored at 3, 24, 48, 72, 96, 120 and 168 h after 177Lu-AB-3PRGD2 administration with serial whole body planar and SPECT/CT imaging (72 or 96h). Analyze and calculate the internal radiation dose of 177Lu-AB-3PRGD2 and evaluate its therapeutic efficiency and response.

ELIGIBILITY:
Inclusion Criteria:

* patients with clear pathological diagnosis and ineffective or progressing clinical conventional treatment;
* tumor lesions with high RGD untake confirmed on 68Ga-RGD PET/CT within one week before the injection of 177Lu-AB-3PRGD2;
* signed written consent.

Exclusion Criteria:

* the exclusion criteria were a serum creatinine level of more than 150 μmol per liter, a hemoglobin level of less than 10.0 g/dl, a white-cell count of less than 4.0× 109/L, a platelet count of less than 100 × 109/L, a total bilirubin level of more than 3 times the upper limit of the normal range and a serum albumin level of more than 3.0 g per deciliter, cardiac insufficiency including carcinoid heart valve disease, a severe allergy or hypersensitivity to radiographic contrast material, claustrophobia;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
StandarStandardized uptake value of 177Lu-AB-3PRGD2 in normal organs and tumors. | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value at each time point in normal organs and tumors will be measured.

SECONDARY OUTCOMES:
Adverse events collection | 2 months
  Adverse events within 2 months after the injection and scanning of patients will be followed and assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China